CLINICAL TRIAL: NCT04661917
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Assess the Efficacy and Safety of BAY 2327949 in Patients With Chronic Kidney Disease (eGFR Range From 25 to 60 mL/Min/1.73 m²) Due to Type 2 Diabetes or Hypertension and at Least One Cardiovascular Comorbidity
Brief Title: A Trial to Learn More About How BAY2327949 Works and How Safe it is in Patients Whose Kidneys Are Damaged Due to High Blood Sugar Levels or High Blood Pressures, and With a Further Disease of the Heart or the Blood Vessels.
Acronym: ASSESS-CKD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn due to company decision
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19225; 2020-002192-35 (EudraCT Number)
Record Dates: First submitted 2020-11-20; First posted 2020-12-10 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Chronic Kidney Disease; Diabetic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY2327949 (Experimental): Participants will receive 60 mg of BAY2327949 (2 tablets of 30 mg) once daily for 28 days.
  Interventions: Drug: BAY2327949
- Placebo (Placebo Comparator): Participants will receive matching placebo once daily for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY2327949 — 60 mg of BAY2327949 (2 tablets of 30 mg, orally) once daily for 28 days.
  Arms: BAY2327949
Drug: Placebo — Matching placebo orally once daily for 28 days.
  Arms: Placebo

SUMMARY:
In people with type 2 diabetes (T2D), the body makes insulin, but cannot use it well. This results in high blood sugar levels causing damage to the blood vessels inside the kidneys.

High blood pressure is a common condition that can cause damage to the blood vessels and heart if it is untreated. High blood pressure is also known as hypertension.

Patients with type 2 diabetes (T2D) or high blood pressure are at a higher risk of having chronic kidney disease (CKD). In people with CKD, the kidneys become damaged and do not work as they should. Over time, the function of the kidney declines more, and this can lead to the requirement for dialysis or kidney transplantation. Most people with CKD are also at risk of heart conditions, such as heart attack or stroke.

In this trial, the researchers want to learn if BAY2327949 reduces the amount of protein in the participants' urine. Protein in the urine is one of the signs of CKD. The researchers will compare the effects of BAY2327949 to a placebo. A placebo looks like the study drug but does not have any medicine in it. BAY2327949 is assumed to increase the blood flow through the kidneys, which may slow down the worsening of the disease. The researchers will use a placebo to learn if the changes seen in the participants are due to BAY2327949 or if the results could be due to chance.

This trial will include about 120 men and women over the age of 45 who have CKD. The participants will have T2D or high blood pressure, and a further disease of the heart or blood vessels.

During the trial, the participants will take either BAY2327949 or a placebo once a day for 28 days. The participants will visit their trial site about 9 times during the trial, and need to provide urine samples to check the participants' CKD symptoms. At the visits, the doctors will ask them if they have any health problems. They will also take blood samples to perform laboratory assessments.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of chronic kidney disease (CKD) with estimated glomerular filtration rate (eGFR) ≥ 25 mL/min/1.73 m^2 but ≤ 60 mL/min/1.73 m^2 (estimated using the CKD-EPI [Epidemiology Collaboration] equation) as assessed during Visit 1, and albuminuria (as measured by urine albumin-to-creatinine ratio [UACR]) in the range of ≥ 30 but ≤ 3000 mg/g, based on the first assessment for Visit 1.
* CKD with a clinical cause of either T2D or hypertension: -- if T2D is the clinical cause, history of type 2 diabetes mellitus as defined by the American Diabetes Association (on treatment with glucose-lowering medications and/or insulin) for at least 2 years before randomization and on a stable therapy with sodium-glucose transport protein 2 (SGLT2) inhibitor for at least 3 months before randomization; -- if hypertension is the clinical cause, patients must have a history of systolic blood pressure (BP) values ≥ 140 mmHg and/or diastolic BP values ≥ 90 mmHg, and on hypertension medication for at least 5 years before randomization.
* Stable treatment with either angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs) at the maximal tolerated labelled daily dose and otherwise stable antihypertensive treatment both for at least 3 months before randomization. If taking an SGLT2 inhibitor, the participant must be on stable treatment for at least 3 months before randomization without any planned changes in dosing during the study period. All treatments must be expected to remain stable over the study period without any planned dose adjustments.
* Body mass index within the range of 18-38 kg/m^2 as evaluated for Visit 1.
* Male participants must agree to use barrier contraception (condoms). Female participants must be of non-child-bearing potential.

Exclusion Criteria:

* Known non-diabetic or non-hypertensive renal disease (e.g. autosomal dominant polycystic kidney disease or autosomal recessive polycystic kidney disease, bilateral clinically relevant renal artery stenosis, lupus nephritis, or ANCA-associated vasculitis, or any other secondary glomerulonephritis).
* Clinical diagnoses of heart failure and persistent symptoms (NYHA [New York Heart Association] class III - IV), or hospitalization for worsening heart failure in the last 3 months prior to signing the informed consent form (ICF).
* Uncontrolled hypertension indicated by >160 mmHg systolic BP or ≥100 mmHg diastolic BP at Visit 1 or Visit 2 or at any unscheduled visit before randomization.
* History of secondary hypertension (i.e., renal artery stenosis, primary aldosteronism, or pheochromocytoma); stroke, transient ischemic cerebral attack, acute coronary syndrome in the last 3 months prior to signing the ICF.
* Dialysis for acute renal failure within the previous 6 months prior to signing the ICF.
* Renal allograft in place or a scheduled kidney transplant within the next 18 weeks from signing the ICF (being on a waiting list does not exclude the participant).
* Hepatic insufficiency classified as Child-Pugh B or C or other significant liver disease (e.g., acute hepatitis, chronic active hepatitis, cirrhosis as indicated by e.g. AST/ALT >3x ULN).
* Active malignancy. Previous malignancies are allowed if there is a 5-year remission- and treatment-free time before signing the ICF.
* Any surgical or medical condition, which in the opinion of the investigator, may place the participant at higher risk from his/her participation in the study, or is likely to prevent the participant from complying with the requirements of the study or completing the study.
* For participants without diabetes: receiving off-label treatment with an SGLT2 inhibitor.
* Indication for immunosuppressants, receiving cytotoxic therapy, immunosuppressive therapy, or other immunotherapy within 6 months prior to signing ICF.
* Combination use of an ACE inhibitor and ARB within 3 months prior to signing ICF.
* Concomitant therapy with drugs that strongly induce or inhibit CYP3A4 (cytochrome P-450 3A4), or that are inhibitors of P-gp (P-glucoprotein).
* Planned change of concomitant medications or dose adjustments during participation in this study.
* Participation in another clinical study with treatment with another investigational product 90 days prior to signing ICF.
* HbA1c > 11% at Visit 1.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-31 (Estimated); Primary Completion 2022-04-25 (Estimated); Study Completion 2022-05-19 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in urine albumin-to-creatinine ratio (UACR) to the end of treatment (Visit 6) | Baseline and Visit 6 (28 days)

SECONDARY OUTCOMES:
Frequency of treatment-emergent adverse events (TEAEs) | From the first treatment with the study intervention until 7 days after the last dose, up to 5 weeks

CONTACTS AND LOCATIONS:
Locations (36):
- Austria (7):
  - Medizinische Universität Graz, Graz, Styria
  - Konventhospital Barmherzige Brüder Linz, Linz, Upper Austria
  - Landeskrankenhaus Feldkirch, Feldkirch, Vorarlberg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Zentrum f. klinische Studien Dr. Hanusch GmbH, Vienna
  - Universitätsklinikum AKH Wien, Vienna
  - Klinik Hietzing, Vienna
- Denmark (6):
  - Aarhus Universitetshospital, Skejby, Aarhus N
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Regionshospitalet Herning, Herning
  - Nordsjællands Hospital, Hillerød
  - Hvidovre Hospital, Hvidovre
  - Odense Universitetshospital, Odense C
- Finland (5):
  - Health Step Finland Oy, Kuopio
  - Päijät-Hämeen keskussairaala, Lahti
  - Oulun yliopistollinen sairaala, Oulu
  - Seinäjoen keskussairaala, Seinäjoki
  - Turun yliopistollinen keskussairaala, kantasairaala, Turku
- Netherlands (4):
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Albert Schweitzer Ziekenhuis, Locatie Dordwijk, Dordrecht
  - Maxima Medisch Centrum, locatie Eindhoven, Eindhoven
  - Albert Schweitzer Ziekenhuis, locatie Zwijndrecht, Zwijndrecht
- Norway (6):
  - AKTIMED Helse AS, Hamar
  - Sykehuset Innlandet HF Hamar, Hamar
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
  - Skedsmo Medisinske Senter, Skedsmokorset
  - Stavanger Helseforskning AS, Stavanger
  - St. Olavs Hospital HF, Trondheim
- Sweden (5):
  - Carlanderska Sjukhuset, Gothenburg
  - ProbarE, Lund
  - Dalecarlia Clinical Research, Rättvik
  - Center For Diabetes, Academic Specialist Center, Stockholm
  - Akademiska Sjukhuset, Uppsala
- Switzerland (3):
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Inselspital Universitätsspital Bern, Bern

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.